CLINICAL TRIAL: NCT03382080
Title: COMPLETE - a School-based Intervention Project to Improve Psychosocial Learning Environments and Increase Completion of Upper Secondary School in Norway: a Cluster Randomized Controlled Trial
Brief Title: A School-based Intervention Project to Increase Completion of Upper Secondary School in Norway
Acronym: COMPLETE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: Oxford Research (Unknown); Nordland Research Institute (Unknown); Voksne for Barn (Unknown); Bodin Upper Secondary School (Unknown); Troms county (Unknown); Nordland county (Unknown); Sogn og Fjordane county (Unknown); Hordaland County (Other Government)
Responsible Party: Principal Investigator, Torill Bogsnes Larsen, Professor, University of Bergen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20161789
Record Dates: First submitted 2017-11-30; First posted 2017-12-22 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Drop Out; Absence; Academic Achievement/Average Grade; Mental Health
Keywords: randomized controlled trial; drop out; upper secondary school; psychosocial learning environments
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dream School Program (DSP) (Experimental): The Dream School Program is a whole school program, involving staff and students, with the aim of creating learning environments where students are confident and experience a sense of belonging, and where mental health is promoted.
  Interventions: Other: Dream School Program
- DSP and Mental Health Support Team (Experimental): A combination of the universal Dream Schoop Program (see description above) and the selective/indicative intervention Mental Health Support Team which is aimed at specific students at risk of dropping out of upper secondary school. It is a systematization of the student services through
  1. Co-location of services and staff working in services
  2. "One open door" to increase accessibility to the services and staff for students
  3. Focus on the transition from lower to upper secondary school
  4. Close follow-up of students at risk to ensure tailored help to each student
  5. Early intervention and follow up when students starts being absent from school
  Interventions: Other: Dream School Program; Other: Mental Health Support Team
- Control (No Intervention): The control group are upper secondary schools who run classes and the school as usual, and do not introduce new programs similar to the Dream School or Mental Health Support Team during the project period.

INTERVENTIONS:
Other: Dream School Program — The Dream School program is a whole school program, involving staff and students, with the aim of creating learning environments where students are confident and experience a sense of belonging, and where mental health is promoted.
  Other Names: Drømmeskolen (Norwegian name)
  Arms: DSP and Mental Health Support Team; Dream School Program (DSP)
Other: Mental Health Support Team — MHST is also a whole school project but aimed at specific students at risk of dropping out. It is a systematisation of the student services through
  1. Co-location of services and staff working in services
  2. "One open door" to increase accessibility to the services and staff for students
  3. Focus on the transition from lower to upper secondary school
  4. Close follow-up of students at risk to ensure tailored help to each student
  5. Early intervention and follow up when students starts being absent from school This work demands cross- and multidisciplinary collaborations within the MHST, between MHST and school leadership, and between lower and upper secondary schools.
  Other Names: Nærværsteam (Norwegian name)
  Arms: DSP and Mental Health Support Team

SUMMARY:
Drop out from upper secondary school represents a risk for the future health and wellbeing of young people. Strengthening of psychosocial aspects of the learning environment may be an effective strategy to promote completion of upper secondary school. The COMPLETE study is a school based cluster randomized controlled trial (RCT) evaluating two school-based interventions, namely the Dream School Program (DSP) and the Mental Health Support Team (MHST) among 1st grade upper secondary school students in four counties in Norway. The interventions aim to improve psychosocial learning environments and subsequently school achievements and decrease drop-out and absence.

Specifically, the COMPLETE study will

1. Evaluate whether the DSP alone

   1. increases completion
   2. increases presence
   3. improves school achievements
   4. improves mental health and wellbeing
2. Evaluate whether the DSP and the MHST combined

   1. increase completion
   2. increase presence
   3. improve school achievements
   4. improve mental health and wellbeing

   The COMPLETE study will also evaluate the effect of the DSP and MHST combined and the DSP alone against secondary outcomes of school satisfaction and loneliness.
3. Evaluate through a process evaluation whether the interventions were implemented in line with guidelines for each of the interventions, and whether the degree of program fidelity has influenced the effect of the interventions on the primary and secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* School inclusion criteria: not been or currently involved in either of the Dream School Program or the Mental Health Support Team or similar programs or research projects
* Student inclusion criteria: student enrolled at any of the included schools.

Exclusion Criteria:

* Schools previously or currently involved in either of the Dream School Program or the Mental Health Support Team or similar programs or research projects.
* Student exclusion criteria: students with special needs or who are illiterate in Norwegian are excluded from the survey assessment, but included in the interventions.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3500 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2020-02-12 (Actual)

PRIMARY OUTCOMES:
Drop-out | Each participant is assessed after 10 months
  If the student has not complete upper secondary school within five years or if the student quit school and is without any regular activity during the course of the study period, i.e. grade 1-3 of upper secondary school
Drop-out | Each participant is assessed after 22 months
  If the student has not complete upper secondary school within five years or if the student quit school and is without any regular activity during the course of the study period, i.e. grade 1-3 of upper secondary school
Drop-out | Each participant is assessed after 34 months
  If the student has not complete upper secondary school within five years or if the student quit school and is without any regular activity during the course of the study period, i.e. grade 1-3 of upper secondary school
Drop-out | Each participant is assessed after 58 months
  If the student has not complete upper secondary school within five years or if the student quit school and is without any regular activity during the course of the study period, i.e. grade 1-3 of upper secondary school
Absence | Each participant is assessed after 10 months
  Total days and hours absent at closure of first school year in upper secondary school
Absence | Each participant is assessed after 22 months
  Total days and hours absent at closure of second school year in upper secondary school
Absence | Each participant is assessed after 34 months
  Total days and hours absent at closure of third school year in upper secondary school
Academic achievement | Each participant is assessed after 10 months
  Average grade at closure of first school year in upper secondary school
Academic achievement | Each participant is assessed after 22 months
  Average grade at closure of second school year in upper secondary school
Academic achievement | Each participant is assessed after 34 months
  Average grade at closure of third school year in upper secondary school
Change from baseline Mental Health at 6 months | Based on self-report in survey assessment at baseline and 6 months
  Short form of Symptom Check List (SCL-5), on a 4 point Likert scale ranging from Not bothered to Very bothered, with higher values indicating a worse outcome.
Change from baseline Mental Health at 18 months | Based on self-report in survey assessment at baseline and 18 months
  Short form of Symptom Check List (SCL-5), on a 4 point Likert scale ranging from Not bothered to Very bothered, with higher values indicating a worse outcome.
Change from baseline Mental Health at 30 months | Based on self-report in survey assessment at baseline and 30 months
  Short form of Symptom Check List (SCL-5), on a 4 point Likert scale ranging from Not bothered to Very bothered, with higher values indicating a worse outcome.
Change in Mental Wellbeing from baseline at 6 months | Based on self-report in survey assessment at baseline and 6 months
  Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS), on a 5 point Likert scale from None of the time to All of the time, with higher values indicating a better outcome
Change from baseline Mental Wellbeing at 18 months | Based on self-report in survey assessment at baseline and 18 months
  Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS), on a 5 point Likert scale from None of the time to All of the time, with higher values indicating a better outcome

SECONDARY OUTCOMES:
Change from baseline School satisfaction at 6 months | Based on self-report in survey assessment at baseline and 6, 18 and 30 months
  Three items from the School Satisfaction Scale, a subscale of the Multidimensional Student's Life Satisfaction Scale. 5 point Likert scale from Completely disagree to Completely agree, with higher values indicating a better outcome.
Change from baseline School satisfaction at 18 months | Based on self-report in survey assessment at baseline and 18 months
  Three items from the School Satisfaction Scale, a subscale of the Multidimensional Student's Life Satisfaction Scale. 5 point Likert scale from Completely disagree to Completely agree, with higher values indicating a better outcome.
Change from baseline School satisfaction at 30 months | Based on self-report in survey assessment at baseline and 30 months
  Three items from the School Satisfaction Scale, a subscale of the Multidimensional Student's Life Satisfaction Scale. 5 point Likert scale from Completely disagree to Completely agree, with higher values indicating a better outcome.
Change from baseline Loneliness at 6 months | Based on self-report in survey assessment at baseline and 6 months
  Loneliness Scale, 5 point Likert scale from Not at all to To a very high degree with higher values indicating a worse outcome.
Change from baseline Loneliness at 18 months | Based on self-report in survey assessment at baseline and 18 months
  Loneliness Scale, 5 point Likert scale from Not at all to To a very high degree with higher values indicating a worse outcome.
Change from baseline Loneliness at 30 months | Based on self-report in survey assessment at baseline and 30 months
  Loneliness Scale, 5 point Likert scale from Not at all to To a very high degree with higher values indicating a worse outcome.

OTHER OUTCOMES:
Change from baseline Social competence at 6 months | Based on self-report in survey assessment at baseline and 6 months
  Wichstrøm Social Competence Scale, a 4 point Likert scale ranging from Describes me very poorly to Describes me very well, with higher values indicating a better outcome.
Change from baseline Social competence at 30 months | Based on self-report in survey assessment at baseline and 30 months
  Wichstrøm Social Competence Scale, a 4 point Likert scale ranging from Describes me very poorly to Describes me very well, with higher values indicating a better outcome.
Change from baseline Social competence at 18 months | Based on self-report in survey assessment at baseline and 18 months
  Wichstrøm Social Competence Scale, a 4 point Likert scale ranging from Describes me very poorly to Describes me very well, with higher values indicating a better outcome.
Change from baseline Relatedness at 6 months | Based on self-report in survey assessment at baseline and 6 months
  Teacher and Classmate Support Scale, a 5 point Likert scale ranging from Completely disagree to Completely agree, with higher values indicating a better outcome.
Change from baseline Relatedness at 18 months | Based on self-report in survey assessment at baseline and 18 months
  Teacher and Classmate Support Scale, a 5 point Likert scale ranging from Completely disagree to Completely agree, with higher values indicating a better outcome.
Change from baseline Relatedness: support at 30 months | Based on self-report in survey assessment at baseline and 30 months
  Teacher and Classmate Support Scale, a 5 point Likert scale ranging from Completely disagree to Completely agree, with higher values indicating a better outcome.
Change from baseline Relatedness: peer connection at 6 months | Based on self-report in survey assessment at baseline and 6 months
  Positive Youth Development Connection Scale, on a 5 point Likert scale, ranging from Almost never or never true to Always true, with higher values indicating a better outcome.
Change from baseline Peer connection at 18 months | Based on self-report in survey assessment at baseline and 18 months
  Positive Youth Development Connection Scale, on a 5 point Likert scale, ranging from Almost never or never true to Always true, with higher values indicating a better outcome.
Change from baseline Peer connection at 30 months | Based on self-report in survey assessment at baseline and 30 months
  Positive Youth Development Connection Scale, on a 5 point Likert scale, ranging from Almost never or never true to Always true, with higher values indicating a better outcome.
Change from baseline Autonomy support at 6 months | Based on self-report in survey assessment at baseline and 6 months
  Ten items from the Learning Climate Scale, a 5 point Likert scale ranging from Strongly disagree to Strongly agree, with higher values indicating a better outcome.
Change from baseline Autonomy support at 18 months | Based on self-report in survey assessment at baseline and 18 months
  Ten items from the Learning Climate Scale, a 5 point Likert scale ranging from Strongly disagree to Strongly agree, with higher values indicating a better outcome.
Change from baseline Autonomy support at 30 months | Based on self-report in survey assessment at baseline and 30 months
  Ten items from the Learning Climate Scale, a 5 point Likert scale ranging from Strongly disagree to Strongly agree, with higher values indicating a better outcome.
Change from baseline Academic competence at 6 months | Based on self-report in survey assessment at baseline and 6 months
  Academic Self-Efficacy Scale, a 5 point Likert scale ranging from Completely disagree to Completely agree, with higher values indicating a better outcome.
Change from baseline Academic competence at 18 months | Based on self-report in survey assessment at baseline and 18 months
  Academic Self-Efficacy Scale, a 5 point Likert scale ranging from Completely disagree to Completely agree, with higher values indicating a better outcome.
Change from baseline Academic competence at 30 months | Based on self-report in survey assessment at baseline and 30 months
  Academic Self-Efficacy Scale, a 5 point Likert scale ranging from Completely disagree to Completely agree, with higher values indicating a better outcome.
Class climate | Based on self-report in survey assessment at baseline
  Caring Climate Scale, on a 5 point Likert scale, ranging from Strongly disagree to Strongly agree, with higher values indicating a better outcome.
Change from 6 month Class climate at 18 months | Based on self-report in survey assessment at 6 and 18 months
  Caring Climate Scale, on a 5 point Likert scale, ranging from Strongly disagree to Strongly agree, with higher values indicating a better outcome.
Change from 6 month Class climate at 30 months | Based on self-report in survey assessment at 6 and 30 months
  Caring Climate Scale, on a 5 point Likert scale, ranging from Strongly disagree to Strongly agree, with higher values indicating a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Torill B Larsen, PhD, Principal Investigator — University of Bergen

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Larsen T, Urke HB, Holsen I, Anvik CH, Olsen T, Waldahl RH, Antonsen KM, Johnson R, Tobro M, Brastad B, Hansen TB. COMPLETE - a school-based intervention project to increase completion of upper secondary school in Norway: study protocol for a cluster randomized controlled trial. BMC Public Health. 2018 Mar 9;18(1):340. doi: 10.1186/s12889-018-5241-z. PMID 29523124
- See also: COMPLETE project web site — https://complete.w.uib.no/